CLINICAL TRIAL: NCT02479932
Title: A Comparison of Skin to Delivery Time at Exztraperitoneal vs. Transpirational Cesarean
Brief Title: A Comparison of Extraperitoneal Versus Transperitoneal Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ragıp Atakan Al, professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 77-2015
Record Dates: First submitted 2015-06-11; First posted 2015-06-24 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Labor Pain
Keywords: Extra-peritoneal cesarean; Intra-peritoneal cesarean
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extraperitoneal cesarean (Active Comparator)
  Interventions: Other: Extraperitoneal cesarean technique
- Transperitoneal cesarean (Active Comparator)
  Interventions: Other: Transperitoneal cesarean technique

INTERVENTIONS:
Other: Transperitoneal cesarean technique — Pfannenstiel-Kerr technique for laparatomy and uterine entry
  Arms: Transperitoneal cesarean
Other: Extraperitoneal cesarean technique — Pfannenstiel incision, paravesical approach to lower uterine segment extraperitoneally and Kerr incision for uterine entry
  Arms: Extraperitoneal cesarean

SUMMARY:
The aim of study is to compare skin-to-delivery time and postoperative morbidity between extraperitoneal cesarean and transpirational cesarean.

ELIGIBILITY:
Inclusion Criteria:

* elective cesarean
* previous cesarean (<4)
* cesarean for distocia

Exclusion Criteria:

* emergency cesarean ( fetal distress)
* risk of obstetrical bleeding
* maternal coagulation defects
* adnexial mass
* uterin myoma at incision site

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Skin-to-delivery time | 1 minute after delivery

SECONDARY OUTCOMES:
Postoperative pain | 24 and 48 hour after cesarean
  Pain will be measured by VAS
Operation time | Two minutes after surgery
  skin-to-skin operation time
Hemoglobin differences | One hour before cesarean and 48 hours after cesarean
Need for analgesic | 24 and 48 hours after cesarean
  All analgesic given after cesarean at hospital
Nausea | Two minutes and 48 hours after cesarean
  Nausea during surgery and after surgery
Vomiting | Two minutes and 48 hours after cesarean
  Nausea during and after surgery
Thoracic shoulder pain | 48 hours after cesarean
  Thoracic shoulder pain after surgery
Urogenital distress measured by Urogenital Distress Inventory | One hour before cesarean and 24 hours after cesarean
Oral intake | 12 and 24 hours postoperatively
  The percentage of patients who tolerates oral intake. Oral intake will be allowed 4-6 hours after cesarean for extraperitoneal group. For intraperitoneal group it will be allowed when patient passed gas.
Anxiety during surgery | One minute after cesarean
  Intense fear or anxiety during surgery without pain (yes or no)
Pain during surgery | One minutes after surgery
  Abdominal pain during surgery (yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: Yunus E TOPDAGI, MD, Principal Investigator — Ataturk University; Omer E Yapca, MD, Study Director — Ataturk University
Locations (1):
- Atatürk Üniversitesi Araştırma Hastanesi, Erzurum, Turkey (Türkiye)